CLINICAL TRIAL: NCT00567268
Title: Drug Use Investigation Of Gabapen
Brief Title: Drug Use Investigation Of Gabapentin
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A9451163
Record Dates: First submitted 2007-11-16; First posted 2007-12-04 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2015-09

CONDITIONS: Epilepsies, Partial
Keywords: Post-Marketing surveillance
MeSH Terms: conditions — Epilepsies, Partial | interventions — Gabapentin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gabapentin: Patients taking Gabapentin
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — GABAPEN Tablets 200mg, GABAPEN Tablets 300mg, GABAPEN Tablets 400mg. GABAPEN is Brand name in Japan.
  Dosage, frequency: According to Japanese LPD, "Normally, oral gabapentin 600 mg, 3 div., should be given on the first day of administration and an effective dose of 1200mg, 3 div, should be given on day 2. From day 3 on, adults should be maintained on oral gabapentin 1200 mg to 1800 mg, 3 div. Subsequently, the maintenance dose should be suitably adjusted depending on the symptoms (up to a maximum daily dose of 2400 mg)".
  Duration: According to the protocol of A9451163, the duration of the investigation for findings regarding safety and efficacy of a patient is from the first drug administration to the 12 weeks after the first administration.

SUMMARY:
The objective of the this surveillance is to collect information about 1)adverse drug reactions not expected from the LPD (unknown adverse drug reactions), 2) the incidence of adverse drug reactions in this surveillance, and 3) factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Gabapentin should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

Patients need to be taking Gabapentin in order to be enrolled in the surveillance

Exclusion Criteria:

Patients not taking Gabapentin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A9451163 prescribes the Gabapentin
Sampling Method: Probability Sample
Enrollment: 1273 (Actual)
Dates: Start 2007-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451163&StudyName=Drug%20Use%20Investigation%20Of%20Gabapentin

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin 200, 300, 400 mg Tablets: The usual dosage of gabapentin in adults and children aged 13 or older was as follows: oral gabapentin 600 mg, 3 div., was administered on day 1 and an effective dose of 1200 mg, 3 div., was administered on day 2. From day 3 on, oral gabapentin 1200 mg to 1800 mg, 3 div., was administered as the maintenance dose. Subsequently, the maintenance dose was suitably adjusted depending on the symptoms (up to a maximum daily dose of 2400 mg).
Period: Overall Study
Arm/Group | Gabapentin 200, 300, 400 mg Tablets
Started | 1194
Completed | 1144
Not Completed | 50
Not completed — Protocol Violation | 7
Not completed — Lost to Follow-up | 36
Not completed — No Visit After First Day of Treatment | 2
Not completed — No Drug Administration | 4
Not completed — Safety Evaluation "Not Assessable" | 1

BASELINE CHARACTERISTICS:
Population: In total, 1194 participants were enrolled in the study. Of the 1194 participants, a total of 50 participants were excluded from the baseline analysis for the following reasons: protocol violation, lost to follow-up, no visit after first day of treatment, no drug administration, and safety evaluation "Not Assessable".
Arm/Group | Gabapentin 200, 300, 400 mg Tablets
Number analyzed (Participants) | 1144
Age, Customized [Number; unit: participants] — Participants taking gabapentin oral tablets 200, 300, or 400 mg according to the Japanese package insert.
  participants
    <65 years | 1001
    >=65 years | 143
Sex: Female, Male [Count of Participants; unit: Participants] — Participants taking gabapentin oral tablets 200, 300, or 400 mg according to the Japanese package insert.
  Participants
    Female | 542
    Male | 602

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events Unexpected From Japanese Package Insert
Description: A treatment-related adverse event was any untoward medical occurrence attributed to gabapentin in a participant who received gabapentin. Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to gabapentin was assessed by the sponsor (Pfizer Japan Inc.).
Time Frame: 12 weeks
Population: The safety analysis population comprised of participants who had met the inclusion criteria and had taken gabapentin at least once.
Measure: Number; unit: participants
Arm/Group | Gabapentin 200, 300, 400 mg Tablets
Number analyzed (Participants) | 1144
participants | 27

2. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to gabapentin in a participant who received gabapentin. Relatedness to gabapentin was assessed by the sponsor (Pfizer Japan Inc.).
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Gabapentin 200, 300, 400 mg Tablets
Number analyzed (Participants) | 1144
participants | 231

3. Primary Outcome: Clinical Efficacy Rate
Description: Clinical efficacy rate, which was defined as the percentage of participants who achieved clinical efficacy over the total number of efficacy analysis population, was presented along with the corresponding exact 2-sided 95% CI. For the basis of efficacy evaluation, frequencies of epileptic seizure were recorded for the periods during the previous 4 weeks from the treatment start date, and that from the end date of observation (12 weeks after the treatment start date, or date of which treatment was terminated before reaching 12 weeks). Clinical efficacy was assessed according to the following categories: (1) effective, (2) not effective, or (3) not assessable.
Time Frame: 12 weeks
Population: The efficacy analysis population comprised of the participants who had at least one post-baseline efficacy evaluation for the clinical efficacy and seizure frequency within the safety analysis population. Participants who had disease not eligible for the survey were excluded from the efficacy analysis population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gabapentin 200, 300, 400 mg Tablets
Number analyzed (Participants) | 1045
Percentage of participants | 61.1 [58.1 to 64.1]

4. Secondary Outcome: Response Ratio (R Ratio)
Description: Response Ratio (R Ratio) was calculated by the following formula, where B represented the frequency of epileptic seizures during 4 weeks before gabapentin treatment, whereas T represented the frequency of epileptic seizures during 4 weeks at the end of observation period of gabapentin treatment: R Ratio= (T-B) / (T+B). R Ratio was within the range of -1 to +1, and a negative value represented a reduction in the frequency of seizure.
Time Frame: 12 weeks
Population: R ratio analysis population comprised of the participants who calculated R ratio at the start of gabapentin treatment and at the end of monitoring period in the efficacy analysis population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Gabapentin 200, 300, 400 mg Tablets
Number analyzed (Participants) | 956
Ratio | -0.410 (0.4855)

5. Secondary Outcome: Responder Rate
Description: Responder rate, which was defined as the percentage of participants whose R ratio was -0.333 or less, was presented along with the corresponding exact 2-sided 95% CI. R ratio of -0.333 or less corresponded to the decrease of epileptic seizure frequency by 50% or more.
Time Frame: 12 weeks
Population: Responder rate analysis population comprised of the participants who calculated R ratio at the start of gabapentin treatment and at the end of monitoring period in the efficacy analysis population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gabapentin 200, 300, 400 mg Tablets
Number analyzed (Participants) | 956
Percentage of participants | 55.0 [51.8 to 58.2]

6. Secondary Outcome: Percent Reduction From Baseline in Epileptic Seizure Frequency
Description: Percent reduction from the baseline in epileptic seizure frequency, was calculated by the following formula, where B represented the frequency of epileptic seizures during 4 weeks before gabapentin treatment, whereas T represented the frequency of epileptic seizures during 4 weeks at the end of observation period of gabapentin treatment: Reduction from the baseline in epileptic seizure frequency (%) = [(T-B)/B] X 100.
Time Frame: 12 weeks
Population: The analysis population comprised of the participants whose frequency of epileptic seizures during 4 weeks before gabapentin treatment (represented by B) was at least once within the R ratio analysis population.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Gabapentin 200, 300, 400 mg Tablets
Number analyzed (Participants) | 950
Percentage | -34.0 (103.70)

7. Other Pre Specified Outcome: Number of Participants With Treatment-Related Adverse Events by Age Across 7 Categories
Description: A treatment-related adverse event was any untoward medical occurrence attributed to gabapentin in a participant who received gabapentin. Participants with treatment-related adverse events were counted by age across 7 categories to assess whether the age was a risk factor for the treatment-related adverse events.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Age <15 Years: Participants <15 years of age taking gabapentin oral tablets 200, 300, or 400 mg according to the Japanese package insert
- Age >=15 and <25 Years: Participants >=15 and <25 years of age taking gabapentin oral tablets 200, 300, or 400 mg according to the Japanese package insert
- Age >=25 and <35 Years: Participants >=25 and <35 years of age taking gabapentin oral tablets 200, 300, or 400 mg according to the Japanese package insert
- Age >=35 and <45 Years: Participants >=35 and <45 years of age taking gabapentin oral tablets 200, 300, or 400 mg according to the Japanese package insert
- Age >=45 and <55 Years: Participants >=45 and <55 years of age taking gabapentin oral tablets 200, 300, or 400 mg according to the Japanese package insert
- Age >=55 and <65 Years: Participants >=55 and <65 years of age taking gabapentin oral tablets 200, 300, or 400 mg according to the Japanese package insert
- Age >=65 Years: Participants >=65 years years of age taking gabapentin oral tablets 200, 300, or 400 mg according to the Japanese package insert
Arm/Group | Age <15 Years | Age >=15 and <25 Years | Age >=25 and <35 Years | Age >=35 and <45 Years | Age >=45 and <55 Years | Age >=55 and <65 Years | Age >=65 Years
Number analyzed (Participants) | 168 | 189 | 204 | 207 | 106 | 127 | 143
participants | 27 | 31 | 52 | 58 | 15 | 26 | 22
Statistical Analysis 1: Comparison: Age <15 Years vs Age >=15 and <25 Years vs Age >=25 and <35 Years vs Age >=35 and <45 Years vs Age >=45 and <55 Years vs Age >=55 and <65 Years vs Age >=65 Years; The risk factor tested was "age". The null hypothesis was that there was no association between the age and the number of responders to the treatment with gabapentin; Test type: Superiority or Other; p = 0.004, Fisher Exact

8. Other Pre Specified Outcome: Number of Participants With Treatment-Related Adverse Events by Number of Concomitant Antiepileptic Drugs at Baseline
Description: A treatment-related adverse event was any untoward medical occurrence attributed to gabapentin in a participant who received gabapentin. Participants with treatment-related adverse events were counted by the number of concomitant antiepileptic drugs at baseline across 5 categories to assess whether the number of concomitant antiepileptic drugs at baseline was a risk factor for the treatment-related adverse events.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- No Concomitant Antiepileptic Drug: Participants taking no concomitant antiepileptic drug at baseline
- One Concomitant Antiepileptic Drug: Participants taking one concomitant antiepileptic drug at baseline
- Two Concomitant Antiepileptic Drugs: Participants taking two concomitant antiepileptic drugs at baseline
- Three Concomitant Antiepileptic Drugs: Participants taking three concomitant antiepileptic drugs at baseline
- Four or More Concomitant Antiepileptic Drugs: Participants taking four or more concomitant antiepileptic drugs at baseline
Arm/Group | No Concomitant Antiepileptic Drug | One Concomitant Antiepileptic Drug | Two Concomitant Antiepileptic Drugs | Three Concomitant Antiepileptic Drugs | Four or More Concomitant Antiepileptic Drugs
Number analyzed (Participants) | 67 | 453 | 373 | 202 | 49
participants | 12 | 70 | 91 | 41 | 17
Statistical Analysis 1: Comparison: No Concomitant Antiepileptic Drug vs One Concomitant Antiepileptic Drug vs Two Concomitant Antiepileptic Drugs vs Three Concomitant Antiepileptic Drugs vs Four or More Concomitant Antiepileptic Drugs; The risk factor tested was "number of concomitant antiepileptic drugs at baseline". The null hypothesis was that there was no linear trend in the number of responders to the treatment with gabapentin across increasing levels of the number of concomitant antiepileptic drugs at baseline; Test type: Superiority or Other; p = 0.003, Fisher Exact
Statistical Analysis 2: Comparison: No Concomitant Antiepileptic Drug vs One Concomitant Antiepileptic Drug vs Two Concomitant Antiepileptic Drugs vs Three Concomitant Antiepileptic Drugs vs Four or More Concomitant Antiepileptic Drugs; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.003, Cochran-Armitage

9. Other Pre Specified Outcome: Number of Participants Who Responded to Treatment With Gabapentin by Age (<65 Versus >=65 Years)
Description: Participants who responded to the treatment with gabapentin were counted by age (<65 vs. >=65 years) to assess whether the age was a factor affecting the treatment efficacy.
Time Frame: 12 weeks
Population: The efficacy analysis population comprised of the participants who had at least one post-baseline efficacy evaluation for the clinical efficacy and seizure frequency in the safety analysis population. Participants who had diseases not eligible for the survey were excluded from the efficacy analysis population.
Measure: Number; unit: participants
Groups:
- Age <65 Years: Participants <65 years of age who responded to the treatment with gabapentin
- Age >=65 Years: Participants >=65 years of age who responded to the treatment with gabapentin
Arm/Group | Age <65 Years | Age >=65 Years
Number analyzed (Participants) | 933 | 112
participants | 545 | 94
Statistical Analysis 1: Comparison: Age <65 Years vs Age >=65 Years; The factor tested was "age". The null hypothesis was that there was no difference between <65 years and >=65 years in the number of participants who responded to the treatment with gabapentin; Test type: Superiority or Other; p < 0.001, Chi-squared

10. Other Pre Specified Outcome: Number of Participants Who Responded to Treatment With Gabapentin by Age Across 7 Categories
Description: Participants who responded to the treatment with gabapentin were counted by age across 7 categories to assess whether the age was a factor affecting the treatment efficacy.
Time Frame: 12 weeks
Population: as for outcome 9
Measure: Number; unit: participants
Groups:
- Age <15 Years: Participants <15 years of age who responded to the treatment with gabapentin
- Age >=15 and <25 Years: Participants >=15 and <25 years of age who responded to the treatment with gabapentin
- Age >=25 and <35 Years: Participants >=25 and <35 years of age who responded to the treatment with gabapentin
- Age >=35 and <45 Years: Participants >=35 and <45 years of age who responded to the treatment with gabapentin
- Age >=45 and <55 Years: Participants >=45 and <55 years of age who responded to the treatment with gabapentin
- Age >=55 and <65 Years: Participants >=55 and <65 years of age who responded to the treatment with gabapentin
Arm/Group | Age <15 Years | Age >=15 and <25 Years | Age >=25 and <35 Years | Age >=35 and <45 Years | Age >=45 and <55 Years | Age >=55 and <65 Years | Age >=65 Years
Number analyzed (Participants) | 161 | 182 | 188 | 196 | 96 | 110 | 112
participants | 93 | 91 | 102 | 113 | 64 | 82 | 94
Statistical Analysis 1: Comparison: Age <15 Years vs Age >=15 and <25 Years vs Age >=25 and <35 Years vs Age >=35 and <45 Years vs Age >=45 and <55 Years vs Age >=55 and <65 Years vs Age >=65 Years; The factor tested was "age". The null hypothesis was that there was no association between the age and the number of participants who responded to the treatment with gabapentin; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Age <15 Years vs Age >=15 and <25 Years vs Age >=25 and <35 Years vs Age >=35 and <45 Years vs Age >=45 and <55 Years vs Age >=55 and <65 Years vs Age >=65 Years; The factor tested was "age". The null hypothesis was that there was no linear trend in the number of responders to the treatment with gabapentin across increasing levels of age categories; Test type: Superiority or Other; p < 0.001, Cochran-Armitage

11. Other Pre Specified Outcome: Number of Participants Who Responded to Treatment With Gabapentin by Severity of Partial Epileptic Seizure
Description: Participants who responded to the treatment with gabapentin were counted by the severity of partial epileptic seizure (mild, moderate and severe) to assess whether the severity of partial epileptic seizure was a factor affecting the treatment efficacy.
Time Frame: 12 weeks
Population: The efficacy analysis population comprised of the participants who had at least one post-baseline efficacy evaluation for the clinical efficacy and seizure frequency in the safety analysis population. Participants who who had diseases not eligible for the survey were excluded from the efficacy analysis population.
Measure: Number; unit: participants
Groups:
- Mild: Participants with mild epilepsy who responded to the treatment with gabapentin
- Moderate: Participants with moderate epilepsy who responded to the treatment with gabapentin
- Severe: Participants with severe epilepsy who responded to the treatment with gabapentin
Arm/Group | Mild | Moderate | Severe
Number analyzed (Participants) | 220 | 595 | 220
participants | 150 | 363 | 118
Statistical Analysis 1: Comparison: Mild vs Moderate vs Severe; The factor tested was "severity of partial epileptic seizure ". The null hypothesis was that there was no association between the degree of severity of partial epileptic seizure (mild, moderate, and severe) and the number of participants who responded to the treatment with gabapentin; Test type: Superiority or Other; p = 0.008, Chi-squared
Statistical Analysis 2: Comparison: Mild vs Moderate vs Severe; The factor tested was "severity of partial epileptic seizure". The null hypothesis was that there was no linear trend in the number of responders to the treatment with gabapentin across the degree of severity of partial epileptic seizure (mild, moderate, and severe); Test type: Superiority or Other; p = 0.002, Cochran-Armitage

12. Other Pre Specified Outcome: Number of Participants Who Responded to Treatment With Gabapentin by Baseline Frequency of Epileptic Seizure
Description: Participants who responded to the treatment with gabapentin were counted by the baseline frequency of epileptic seizure (<=8 vs. >8 episodes) to assess whether the baseline frequency of epileptic seizure was a factor affecting the treatment efficacy.
Time Frame: 12 weeks
Population: as for outcome 9
Measure: Number; unit: participants
Groups:
- <=8 Episodes: Participants with baseline episodes of epileptic seizure below 8 who responded to the treatment with gabapentin
- >8 Episodes: Participants with baseline episodes of epileptic seizure more than 8 who responded to the treatment with gabapentin
- Unknown: Participants with unknown frequency of baseline episodes who responded to the treatment with gabapentin
Arm/Group | <=8 Episodes | >8 Episodes | Unknown
Number analyzed (Participants) | 688 | 303 | 54
participants | 432 | 166 | 41
Statistical Analysis 1: Comparison: <=8 Episodes vs >8 Episodes; The factor tested was "baseline frequency of epileptic seizure". The null hypothesis was that there was no difference between the baseline frequency of epileptic seizure and the number of participants who responded to the treatment with gabapentin; Test type: Superiority or Other; p = 0.018, Chi-squared

13. Other Pre Specified Outcome: Number of Participants Who Responded to Treatment With Gabapentin by Number of Concomitant Antiepileptic Drugs at Baseline
Description: Participants who responded to the treatment with gabapentin were counted by the number of concomitant epileptic drugs at baseline across 5 categories to assess whether the number of concomitant epileptic drugs at baseline was a factor affecting the treatment efficacy.
Time Frame: 12 weeks
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | No Concomitant Antiepileptic Drug | One Concomitant Antiepileptic Drug | Two Concomitant Antiepileptic Drugs | Three Concomitant Antiepileptic Drugs | Four or More Concomitant Antiepileptic Drugs
Number analyzed (Participants) | 41 | 413 | 357 | 190 | 44
participants | 32 | 295 | 190 | 98 | 24
Statistical Analysis 1: Comparison: No Concomitant Antiepileptic Drug vs One Concomitant Antiepileptic Drug vs Two Concomitant Antiepileptic Drugs vs Three Concomitant Antiepileptic Drugs vs Four or More Concomitant Antiepileptic Drugs; The factor tested was "number of concomitant antiepileptic drugs at baseline". The null hypothesis was that there was no association between the number of concomitant antiepileptic drugs at baseline and the number of participants who responded to the treatment with gabapentin; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: No Concomitant Antiepileptic Drug vs One Concomitant Antiepileptic Drug vs Two Concomitant Antiepileptic Drugs vs Three Concomitant Antiepileptic Drugs vs Four or More Concomitant Antiepileptic Drugs; The factor tested was "number of concomitant antiepileptic drugs at baseline". The null hypothesis was that there was no linear trend in the number of responders to the treatment with gabapentin across increasing levels of the number of concomitant antiepileptic drugs at baseline; Test type: Superiority or Other; p < 0.001, Cochran-Armitage

14. Other Pre Specified Outcome: Number of Participants Who Responded to Treatment With Gabapentin by Baseline Creatinine Clearance
Description: Participants who responded to the treatment with gabapentin were counted by the baseline creatinine clearance (CLcr) across 6 categories to assess whether the baseline CLcr was a factor affecting the treatment efficacy.
Time Frame: 12 weeks
Population: as for outcome 9
Measure: Number; unit: participants
Groups:
- CLcr >=60 mL/Min: Participants with baseline creatinine clearance >=60 mL/min
- CLcr >=30 and <60 mL/Min: Participants with baseline creatinine clearance >=30 and <60 mL/min
- CLcr >=15 and <30 mL/Min: Participants with baseline creatinine clearance >=15 and <30 mL/min
- CLcr >=5 and <15 mL/Min: Participants with baseline creatinine clearance >=5 and <15 mL/min
- CLcr <5 mL/Min: Participants with baseline creatinine clearance <5 mL/min
- Unkown: Participants with unkown baseline creatinine clearance
Arm/Group | CLcr >=60 mL/Min | CLcr >=30 and <60 mL/Min | CLcr >=15 and <30 mL/Min | CLcr >=5 and <15 mL/Min | CLcr <5 mL/Min | Unkown
Number analyzed (Participants) | 439 | 36 | 4 | 1 | 0 | 565
participants | 284 | 28 | 4 | 1 |  | 322
Statistical Analysis 1: Comparison: CLcr >=60 mL/Min vs CLcr >=30 and <60 mL/Min vs CLcr >=15 and <30 mL/Min vs CLcr >=5 and <15 mL/Min vs CLcr <5 mL/Min; The factor tested was "baseline creatinine clearance". The null hypothesis was that there was no linear trend in the number of responders to the treatment with gabapentin across increasing levels of the baseline creatinine clearance; Test type: Superiority or Other; p = 0.025, Cochran-Armitage

15. Other Pre Specified Outcome: Number of Participants Who Responded to Treatment With Gabapentin by Presence or Absence of Non-Drug Therapy
Description: Participants who responded to the treatment with gabapentin were counted by the presence or absence of non-drug therapy to assess whether the non-drug therapy was a factor affecting the treatment efficacy.
Time Frame: 12 weeks
Population: as for outcome 9
Measure: Number; unit: participants
Groups:
- Presence of Non-Drug Therapy: Participants with non-drug therapy who responded to treatment with gabapentin
- Absence of Non-Drug Therapy: Participants without non-drug therapy who responded to treatment with gabapentin
Arm/Group | Presence of Non-Drug Therapy | Absence of Non-Drug Therapy
Number analyzed (Participants) | 45 | 1000
participants | 34 | 605
Statistical Analysis 1: Comparison: Presence of Non-Drug Therapy vs Absence of Non-Drug Therapy; The factor tested was "non-drug therapy". The null hypothesis was that there was no difference between the non-drug therapy and the number of participants who responded to the treatment with gabapentin; Test type: Superiority or Other; p = 0.043, Chi-squared

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The frequency of adverse events. The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Gabapentin 200, 300, 400 mg Tablets
Serious Adverse Events (participants affected / at risk) | 29/1144
Other Adverse Events (participants affected / at risk) | 248/1144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin 200, 300, 400 mg Tablets (N=1144)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2)
Vogt-Koyanagi-Harada syndrome (Eye disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.50% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin 200, 300, 400 mg Tablets (N=1144)
Decreased activity (Psychiatric disorders) | 8 (8)
Ataxia (Nervous system disorders) | 6 (6)
Somnolence (Nervous system disorders) | 137 (137)
Headache (Nervous system disorders) | 6 (6)
Dizziness (Nervous system disorders) | 40 (40)
Hepatic function abnormal (Hepatobiliary disorders) | 6 (6)
Malaise (General disorders) | 8 (8)
Gamma-glutamyltransferase increased (Investigations) | 11 (11)
White blood cell count decreased (Investigations) | 7 (7)
Nausea (Gastrointestinal disorders) | 6 (6)
Convulsion (Nervous system disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.